CLINICAL TRIAL: NCT03446066
Title: Cognitive Assessment in Excessive Daytime Sleepiness: Electrophysiological Study.
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Leqaa El Mekkawy, assistant lecturer, Kasr El Aini Hospital
Other Study IDs: 23101985
Record Dates: First submitted 2018-01-28; First posted 2018-02-26 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- case group: 20 cases suffering from excessive daytime sleepiness (4 females and 16 males) with their age range 32-58yrs and BMI range is 24.97-39.06 kg/m2
- control group: 20 healthy subjects (5 females and 15 males) with their age range 31-55yrs and BMI range is 23.40-43.0 kg/m2

SUMMARY:
Cognition was assessed using Minimental state examination (MMSE), Trail making tests A and B (TMT) tests, P300 and quantitative electroencephalography (QEEG) sleepiness was assessed using Epworth Sleepiness Scale (ESS), Karolinska sleepiness scale (KSS) and QEEG also polysomnography (PSG) was done for all participated subjects

DETAILED DESCRIPTION:
*The study is a case control study included 40 subjects, divided into 20 cases suffering from Excessive daytime sleepiness and 20 healthy control group.

all participants were subjected to:

1. Careful history taking and Complete neurological examination.
2. Initial assessment of cognition and sleepiness by two scales which were done once before sleep: Epworth Sleepiness Scale (ESS) and Minimental state examination (MMSE)
3. Scales and neurophysiological studies done before and after sleep:Karolinska sleepiness scale (KSS), Trail making tests A and B (TMT), P300, and QEEG
4. Polysomnography (PSG)

   * EEG was recorded for 20 minutes duration before and after sleep recording. In each EEG recording, alpha attenuation test (AAT) was done after 10 minutes of recording basal resting EEG, then the absolute power of 5 electrodes (CZ, T3, T4, T5, T6,) were studied in the following frequency bands: delta (0.5-3Hz), theta (4-7 Hz) and also the absolute power of (O1, O2) were studied in delta, theta and alpha (8-12 Hz) bands.

ELIGIBILITY:
Inclusion Criteria:

* The age ranges from 18 to 60 years. The age of all included subjects was 31-58 yrs old.
* The body mass index (BMI) range is 24.97-39.06 kg/m2 in patients and 23.40-43.0 kg/m2 in control group.
* Patients suffering from excessive daytime sleepiness symptoms according to the International Classification of Sleep Disorders definitions.

Exclusion Criteria:

* Patients suffering from EDS secondary to any sleep disorder other than sleep disordered breathing.
* Chronic debilitating disease as diabetes mellitus , hypertension or hyper- or hypo-thyroidism.
* Medications that could affect attention or vigilance as Benzodizipines, anti-psychotics or anti-epileptics.

Ages: 31 Years to 58 Years | Sex: All
Age Groups: Adult
Study Population: 20 patients suffering from EDS 20 healthy subgects
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-12-23 (Actual)

PRIMARY OUTCOMES:
change in Quantitative electroencephalography (QEEG) and P300 results from before to after single night sleep record in patients with excessive daytime sleepiness (EDS) | 1 year
  the results of QEEG and P300 in patients with EDS before and after sleep

SECONDARY OUTCOMES:
potential integration of quantitative EEG and P300 as diagnostic tools for cognition and EDS. | 1year
  usage of electrophysiological tools for diagnosis of cognitive affection and sleepiness in EDS patients

CONTACTS AND LOCATIONS:
Overall Officials: Mona Nada, prof., Study Director — Cairo University